CLINICAL TRIAL: NCT04502589
Title: Open Label Pilot Study of Perampanel for the Treatment of Alcohol Use Disorder
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM20015846; R21AA026681 (NIH)
Record Dates: First submitted 2020-08-04; First posted 2020-08-06 (Actual); Results first posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Alcohol Disorders
MeSH Terms: conditions — Alcohol-Related Disorders | interventions — perampanel; Disulfiram

STUDY DESIGN:
Intervention Model Description: 20 subjects with AUD will be randomized 1:1 to one of two groups; perampanel by itself, and perampanel combined with disulfiram.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- perampanel by itself (Active Comparator)
  Interventions: Drug: Perampanel Tablet
- Perapanel with Disulfiram (Active Comparator)
  Interventions: Drug: Perampanel Tablet; Drug: Disulfiram

INTERVENTIONS:
Drug: Perampanel Tablet — Subjects will be titrated over 3 weeks to a target dose of 8mg perampanel daily in both groups
Drug: Disulfiram — Disulfiram will be kept at 250mg daily
  Arms: Perapanel with Disulfiram

SUMMARY:
The purpose of this research study is to test the safety, tolerability, and effectiveness of the drug Perampanel when used in persons who drink and wish to stop drinking. Perampanel has been approved by the U.S. Food and Drug Administration (FDA) for the treatment of seizures but has not yet been approved to treat alcohol use disorders. For this reason, it is considered an investigational drug. Some people in this study will receive Perampanel alone and some people will receive Perampanel and Disulfiram, this will be determined by the pharmacy.

DETAILED DESCRIPTION:
Participants will be asked to take a medication (Perampanel or Perampanel + Disulfiram) every day for approximately 8 weeks and have weekly study visits. At these visits, participants will be asked questions about their medical history, drinking behavior and life events, have bloodwork checked routinely, have regular medication counseling, and perform some computer tasks. Throughout the study, there will be regular phone calls from staff. Participants will also be asked to use a device called "Soberlink" which is like an at-home breathalyzer test to help track progress throughout the study.

Participants will be randomly assigned (like the flip of a coin) to receive either Perampanel alone or Peramanel and Disulfiram.

Participation in this study will last up to 10 weeks. Approximately 20 individuals will participate in this study.

This study will sequence all or part of participant's DNA. This is a necessary part of the study.

Before starting the study, participants may be referred to an alcohol detoxification program (medical treatment of an alcoholic), if clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ages 21-70 with DSM-5 AUD;
2. regular heavy drinkers as defined by averaging ≥ 2 heavy drinking days per week over the 60 days baseline pre-treatment TLFB, and recognize a need to completely stop drinking;
3. willingness to provide written, informed consent to participate in the study;
4. Individuals with LFTs that are no more than 2-3 times above the normal levels and with a Child-Pugh score of no greater than 5 will be included and
5. women of child-bearing potential (i.e., no hysterectomy, bilateral oophorectomy, or tubal ligation or <2 years postmenopausal), must be non-lactating, practicing a reliable method of birth control, and have a negative serum pregnancy test prior to initiation of treatment.

Exclusion Criteria:

1. a current, clinically significant physical disease [i.e., neurologic, renal, pulmonary, cardiovascular, hepatic] on the basis of medical history, physical examination, or routine laboratory evaluation that, in the context of the study would represent a risk to the subject, or significant laboratory abnormalities related to hepatic function such as marked elevations of hepatic aminotransferase levels (i.e., AST and ALT) or direct bilirubin;
2. history of renal compromise or current renal disease (as evidenced by serum creatinine above our laboratory's reference limit of 1.7 mg/dL;
3. history of seizure disorder;
4. use of any of a number of medications that might prominently influence drinking patterns or cause risk of harm or injury (e.g., other anticonvulsants, medications to treat AUD, opioid pain medication), currently taking CNS depressants (e.g. benzodiazepines, barbiturates, sedating antihistamines;
5. schizophrenia, bipolar disorder, current major depressive episode, or substantial suicide or violence risk on the basis of history or psychiatric examination;
6. currently dependent on stimulants, opioids or sedatives;
7. subjects with any substantial alcohol withdrawal will be required to be detoxified by regular clinical services prior to study entry;
8. are currently taking any medication that is a moderate to strong CYP3A4 inhibitor or inducer if participants are required to initiate these medications by an outside provider during the course of this study, they will be tapered off the study regimen and we will have them terminate early)
9. are taking phenytoin or warfarin

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-08-11 (Actual); Study Completion 2021-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Arias, MD, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University Inst. for Drug and Alcohol Studies, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Perampanel by Itself | Perapanel With Disulfiram
Started | 2 | 2
Completed | 1 | 2
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Perampanel by Itself | Perapanel With Disulfiram | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percent Abstinent Days
Description: Participant will report the number of alcoholic drinks they consumed during the previous weeks period. Participants will be accessed for the full 12 week titration plus treatment period. However, for the purposes of the study, the percent of days the participant was abstinent will be calculated and reported only for the 8 week active treatment period.
Time Frame: End of treatment, up to 12 weeks
Measure: Mean (Full Range); unit: Percentage of days
Arm/Group | Perampanel by Itself | Perapanel With Disulfiram
Number analyzed (Participants) | 2 | 2
Percentage of days | 3.13 [0 to 6.25] | 100 [100 to 100]

2. Secondary Outcome: Change in Alcohol Craving
Description: Alcohol craving will be assessed using the Alcohol Urge Questionnaire (AUG). The AUG is an 8-item survey asking participants to rate their craving for alcohol on a 1 to 7 scale. The answers are summed yielding a score ranging from 7 to 56 with higher scores indicated higher alcohol craving.
Time Frame: Baseline to end of treatment, up to 12 weeks
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Perampanel by Itself | Perapanel With Disulfiram
Number analyzed (Participants) | 2 | 2
score on a scale | 4 [2 to 6] | -1 [-2 to 0]

3. Secondary Outcome: Percent Heavy Drinking Days
Description: Participant will report the number of alcoholic drinks they consumed during the previous weeks period. Based on participant report, the percent of days the participant drank heavily will be calculated over the 8 week active treatment period.
Time Frame: End of treatment, Up to 8 weeks
Measure: Mean (Full Range); unit: percentage of days
Arm/Group | Perampanel by Itself | Perapanel With Disulfiram
Number analyzed (Participants) | 2 | 2
percentage of days | 73.60 [65.6 to 81.6] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: At baseline and weekly for eight weeks
Description: The Systematic Assessment for Treatment Emergent Events (SAFTEE) is a NIAAA developed assessment for adverse events in alcohol pharmacotherapy trials. The assessment was modified to assess for known side effects of perampanel.
Arm/Group | Perampanel by Itself | Perapanel With Disulfiram
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/2
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Perampanel by Itself (N=2) | Perapanel With Disulfiram (N=2)
Vehicle accident (General disorders) | 1 (1) | 0 (0) — Vehicle accident due to Drowsiness without injury
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Perampanel by Itself (N=2) | Perapanel With Disulfiram (N=2)
Aggression/Anger (Psychiatric disorders) | 2 (3) | 0 (0)
Agitation (Psychiatric disorders) | 2 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (2)
Breathing Diffuculties (General disorders) | 1 (3) | 0 (0)
Confusion/Slow Thinking (Psychiatric disorders) | 2 (4) | 1 (2)
Decreased Coordination (Nervous system disorders) | 1 (3) | 1 (2)
Depressed Mood (Psychiatric disorders) | 1 (1) | 1 (1)
Dizziness (Ear and labyrinth disorders) | 1 (3) | 1 (1)
Double Vision (Eye disorders) | 1 (2) | 1 (1)
Drowsiness (General disorders) | 2 (5) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 2 (2) | 1 (2)
Fatigue (General disorders) | 2 (5) | 2 (4)
Hostility (Psychiatric disorders) | 2 (2) | 2 (4)
Irregular Heartbeat (Cardiac disorders) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 1 (1) | 1 (1)
Itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Lightheadedness (General disorders) | 1 (4) | 1 (1)
Loss of Appetite (Gastrointestinal disorders) | 1 (1) | 0 (0)
Loss of Balance (General disorders) | 1 (3) | 1 (2)
Nausea/Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Panic Attacks (Psychiatric disorders) | 1 (1) | 1 (1)
Restlessness (Psychiatric disorders) | 2 (2) | 0 (0)
Shortness of Breath (General disorders) | 1 (2) | 0 (0)
Speech Problems (Psychiatric disorders) | 1 (2) | 1 (1)
Trouble Speaking or Swallowing (Nervous system disorders) | 1 (2) | 1 (1)
Unsteady Walking (General disorders) | 1 (1) | 1 (2)
Unusual Skin Sensations (Nervous system disorders) | 1 (1) | 2 (2)
Weakness (General disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/89/NCT04502589/Prot_SAP_002.pdf
  • Informed Consent Form (2021-08-10): https://cdn.clinicaltrials.gov/large-docs/89/NCT04502589/ICF_000.pdf